CLINICAL TRIAL: NCT00957957
Title: Gut Hormone Profiling in Peripheral Blood After Bariatric Surgery in Obese Patients With Type 2 Diabetes
Brief Title: Gut Hormone Profiling in Obese Patients With Type 2 Diabetes (MK-0000-134)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0000-134; 2009_002 (Other: Merck)
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Obesity, Morbid; Diabetes Mellitus Type 2
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Participants having elective Roux-en-Y gastric bypass surgery (RYGBP)
- 2: Participants having elective gastric banding surgery (GB)

SUMMARY:
This study will examine changes in various gut-derived hormones in obese type 2 diabetic patients before and after elective bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Documented type 2 diabetes with total disease duration ≤10 years
* BMI of at least 35 kg/m^2
* Patient is a surgical candidate for either RYGBP, GBS or vertical sleeve gastrectomy (VSG)

Exclusion Criteria:

* Any illness that might confound the results of the study or pose additional risk to the patient by participation
* History of stroke, seizures, or other major neurological disorder
* History of cancer
* Patient uses or has used any medication that can alter body weight
* Patient is unwilling or unable to follow study procedures

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Morbidly obese type 2 diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in PYY (Peptide YY) measured by ELISA 4 weeks after RYGBP | Baseline and Week 4

SECONDARY OUTCOMES:
Change from baseline in PYY measured by dMS 4 weeks after RYGBP | Baseline and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Shankar SS, Mixson LA, Chakravarthy M, Chisholm R, Acton AJ, Jones R, Mattar SG, Miller DL, Petry L, Beals CR, Stoch SA, Kelley DE, Considine RV. Metabolic improvements following Roux-en-Y surgery assessed by solid meal test in subjects with short duration type 2 diabetes. BMC Obes. 2017 Mar 1;4:10. doi: 10.1186/s40608-017-0149-1. eCollection 2017. PMID 28265415